CLINICAL TRIAL: NCT07361536
Title: Cardiovascular Structure and Function in Mucopolysaccharidosis Types I and IVA
Brief Title: Cardiac Structure and Function in MPS
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13984001; 1R01HL173371-01A1 (NIH)
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: MPS I; MPS IV A; MPS - Mucopolysaccharidosis; MPS IVA
Keywords: mucopolysaccharidosis; carotid; cardiovascular; biomarker; observational
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Plasma
  * Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MPS: Participants diagnosed with MPS I or MPS IVA
- Control: Participants who do not have an MPS diagnosis

SUMMARY:
The purpose of this study is to better understand how heart and blood vessel problems develop in people with Mucopolysaccharidosis (MPS). The investigators are looking at certain substances in the body called GAGs and proteoglycans to see how they affect the heart. The investigators also want to find reliable blood and urine markers that can help us track heart health and guide future treatments.

This study aims to answer two main questions:

1. Do people with MPS show faster changes in their blood vessels over time (such as thickening or stiffening of the carotid artery) compared to people without MPS?
2. Do people with MPS have higher levels of certain proteins in their blood (such as clusterin and inflammatory markers) that are linked to blood vessel changes?

What participants will do?

Participants will complete the following tests once a year for 4 years:

* Carotid ultrasound: an imaging test that looks at the blood vessels in the neck.
* Echocardiogram: an ultrasound of the heart.
* Blood draw
* Urine collection

These tests help the investigators track changes in heart and blood vessel health over time.

ELIGIBILITY:
Inclusion Criteria:

1. Any Participant with a molecularly confirmed diagnosis of mucopolysaccharidosis is eligible to enroll in this study
2. Any healthy participant without a diagnosis of mucopolysaccharidosis whose age and biological sex can be matched with an enrolled mucopolysaccharidosis participant
3. Parental / patient informed consent

Exclusion Criteria:

1. Any reason that the investigators would deem a patient not eligible to participate in this study
2. Inability to participate in the assessments required for this study

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be drawn from each participating site's existing patient population. Eligible individuals who meet protocol-defined criteria and are willing to take part in annual study visits will be invited to enroll. The study population will therefore consist of patients receiving care at the participating institutions who consent to ongoing observational follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac and Carotid Structure and Function | Year 1, Year 2, Year 3, and Year 4
  1) We aim to annually assess cardiac and carotid structure and function utilizing ultrasonography, in participants with mucopolysaccharidoses and matched control participants

SECONDARY OUTCOMES:
Measure biomarkers | Year 1, Year 2, Year 3, and Year 4
  2) We aim to annually measure circulating levels of clusterin, elastin, cathepsin S, and cytokines in participants with mucopolysaccharidoses and matched control participants

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children'S Hospital of Orange County, Orange, California
  - University of Minnesota, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri